CLINICAL TRIAL: NCT03839979
Title: Association Between HCV Viral Hepatitis, Blood Sugar Level and Systolic Blood Pressure in the Egyptian Population
Brief Title: HCV Viral Hepatitis, Blood Sugar Level and Systolic Blood Pressure in Egypt
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Wageh Mohareb, Principal Investigator, Cairo University
Other Study IDs: One million healthy citizen 18
Record Dates: First submitted 2019-02-09; First posted 2019-02-15 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Hepatitis C, Acute; Diabetes; Hypertension
MeSH Terms: conditions — Hepatitis C; Diabetes Mellitus; Hypertension | interventions — Blood Pressure Determination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- HCV positive patients: Patients tested positive for the hepatitis c virus antibodies by BIOLINE HCV kits.
  Interventions: Diagnostic Test: BIOLINE HCV kits; Diagnostic Test: ACCU-CHEK kits; Diagnostic Test: ErKameter 3000 mercury manometer
- HCV negative patients: Patients tested negative for the hepatitis c virus antibodies by BIOLINE HCV kits.
  Interventions: Diagnostic Test: BIOLINE HCV kits; Diagnostic Test: ACCU-CHEK kits; Diagnostic Test: ErKameter 3000 mercury manometer

INTERVENTIONS:
Diagnostic Test: BIOLINE HCV kits — We used BIOLINE HCV kits to detect the presence of HCV antibodies in stick blood samples of all recruited patients.
  Other Names: diagnosis of viral hepatitis C
Diagnostic Test: ACCU-CHEK kits — For all patients, we measured random blood sugar levels by stick blood samples using ACCU-CHEK kits.
  Other Names: measurement of blood sugar level
Diagnostic Test: ErKameter 3000 mercury manometer — For all patients, we measured systolic blood pressure using ErKameter 3000 mercury manometer.
  Other Names: blood pressure measurement

SUMMARY:
An observational double-blind cohort study that examined the association between HCV viral hepatitis, blood sugar level and systolic blood pressure in the Egyptian population

DETAILED DESCRIPTION:
a cohort study on greater than 70000 Egyptian patients had been conducted. for all patients,1- we detected the Hepatitis C Virus (HCV) RNA antigens ( hepatitis C virus)presence using BIOLINE HCV kits( qualitative test for diagnosis of hepatitis C virus in the blood), For all positive patients, confirmatory rapid screening test was performed and all patients who tested positive twice underwent a qPCR test using QIAampMinElute Virus Spin kit (Thermo Fisher Scientific, Waltham, MA, USA) performed according to the manufacturer's recommended protocol.

2- Investigators measured blood sugar levels for each patient using ACCU-CHEK kits(finger stick sugar level measurement) 3- Measured systolic blood pressure for each patient was measured using mercury meters.

4-for all patients investigators obtained full medical history regarding the presence or absence of chronic diabetes, chronic hypertension, coronary artery disease, kidney impairment with dialysis or chronic obstructive pulmonary disease.

5- for all patients investigators listed age, gender, and body mass index. 66121 patients were negative for HCV and 4852 were positive for HCV. Investigators measured the association between HCV presence, high blood sugar levels and high systolic blood pressure.

It is supposed that this is the largest study in the world that examined both associations.

In a word, this study was responding to a specific question: is hepatitis c virus presence is associated with high blood pressure or high sugar level or both or not associated???

ELIGIBILITY:
Inclusion Criteria

* Egyptian citizens from 18 years to 80 years.

Exclusion Criteria:

* Patients younger than 18 years or older than 80 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Egyptian patients aged 18-80 years.
Sampling Method: Non-Probability Sample
Enrollment: 71975 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
HCV diagnosis | 20 minutes
  Detection of patients who are HCV positive or negative
Measurement of blood sugar level in mg/dl | 1 minute
  Detection of the percentage of patients with high blood sugar level in HCV positive or negative patients
Measurement of systolic blood pressure in mmHg | 1 minute
  Detection of the percentage of patients with high systolic blood pressure in HCV positive or negative patients

CONTACTS AND LOCATIONS:
Locations (1):
- Egyptian Ministry of Health, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared with other researchers.